CLINICAL TRIAL: NCT06493721
Title: Clear Aligner Treatment for Upper Incisor Crowding With Low-Level Laser Therapy: A Comparative Clinical Study
Brief Title: Clear Aligner Treatment With and Without Low Level Laser Therapy for Upper Incisor Crowding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Nada Ashraf Ali, Demonstrator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHO-109-2-M
Record Dates: First submitted 2024-06-29; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Crowding of Anterior Maxillary Teeth
Keywords: Clear aligner treatment; Low level laser therapy; Clear aligner therapy; Accelerated orthodontics; orthodontic tooth movement; upper incisor crowding; orthodontic pain
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clear aligner only (Experimental): Clear aligner therapy group only
  Interventions: Procedure: Clear Aligner Treatment
- Low level laser (Experimental): Clear aligner therapy with low level laser therapy
  Interventions: Procedure: Clear Aligner Treatment; Procedure: Low level laser

INTERVENTIONS:
Procedure: Clear Aligner Treatment — Clear aligner therapy to treat incisors crowding
Procedure: Low level laser — Apply clear aligner therapy with low level laser application on incisors
  Arms: Low level laser

SUMMARY:
The goal of this clinical trial is to assess the effect of Low Level Laser Therapy (LLLT) on Upper Incisor Crowding using Clear Aligner Treatment (CAT).

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the effect of Low Level Laser Therapy (LLLT) on Upper Incisor Crowding using Clear Aligner Treatment (CAT) on healthy patients (16-23 years old) with complete set of dentition and Angle class I. The main questions to answer are:

1. Evaluate rate of Upper Incisor Decrowding using CAT and LLLT
2. Does LLLT affect pain during CAT?

Researchers will compare CAT with LLLT to CAT without LLLT to see if the LLLT will accelerate Orthodontic Tooth Movement.

Participants will:

* Change to a new aligner every 7 days.
* Visit the clinic every week for checkup.
* Log in pain scores every 6, 24, 48 and 72 hours after delivery of new aligners.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age ranging from 16-23 years old with Angle class I malocclusion and upper anterior crowding.
2. Healthy, compliant and internally motivated patient.
3. Full set of maxillary permanent dentition except third molar.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. Any systemic diseases that could interfere with orthodontic treatment.
3. Gross gingival or periodontal problems

Ages: 16 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Rate of tooth movement | Initial alignment at the end of 3rd month during treatment planning of clear aligner
  Calculate rate of anterior incisor decrowding using digital measurement in millimetre

SECONDARY OUTCOMES:
Pain level | Initial alignment at the end of 3rd month phase during treatment planning of clear aligner
  Will Low Level Laser Therapy decrease pain levels during clear aligner treatment. Evaluated using Numerical Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Samir Abdo, Study Director — Faculty of Dental Medicine, Girls Branch, Al Azhar University
Locations (1):
- Faculty of Dental Medicine for Girls Al-Azhar University, Cairo, Egypt